CLINICAL TRIAL: NCT02649699
Title: Quantitative and Multi-Parametric 3D Magnetic Resonance Imaging of Primary Brain Tumors
Brief Title: Multi-Parametric Brain Cancer MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREBA CC 14-0163
Record Dates: First submitted 2015-12-31; First posted 2016-01-07 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Brain Tumors
Keywords: Primary Brain Cancer
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Additional 3D MRI scans (Other): Participating patients will receive additional 3D MRI scans during pre and post RT planning for their primary brain tumors.
  Interventions: Other: 3D MRI Scans

INTERVENTIONS:
Other: 3D MRI Scans — Patients will receive additional MRI scans before commencing their radiation treatment, at 3-4 months, 6 months and 12 months post RT as well as at recurrence or suspected recurrence.

SUMMARY:
The purpose of this pilot study is to test new magnetic resonance imaging (MRI) acquisition and processing techniques on primary brain tumor patients. The objectives are to improve image-guided radiation therapy (IGRT) planning (first part of the study) and treatment monitoring (second part).

DETAILED DESCRIPTION:
In traditional IGRT the radiation treatment is planned and simulated on computers using x-ray computed tomography (CT) images alone or a combination of CT and MRI. The CT mostly provides information about attenuation of radiation beams needed for the dose simulations because most tumours are more readily identified and contoured with MRI. However, fusion of CT and MR images is prone to error and is a time-consuming process that cannot be automated reliably. Previous research (Stanescu et al.) has shown that the attenuation information can be obtained from MRI which, unlike CT, does not use ionizing radiation to create images. Eliminating the CT scan is therefore possible and beneficial to both the patient, who avoids an additional dose of diagnostic x rays, and to the health care system which saves resources that can be used elsewhere.

Our new MRI acquisition and processing techniques (performed at 3 tesla i.e. 3T) enable:

1. the extraction of 4 different quantitative parameters (hence "multi-parametric MRI", quantitative MRI or relaxometry) that are normally not accessible in traditional MRI, and
2. the automatic classification of tissues (e.g. bone, air, adipose, soft tissue, etc.) which is needed for dose computation in IGRT planning

In the first part of the study (dosimetry) these MRI methods will be used to generate a pseudo-CT to replace the traditional CT data. The hypothesis is that dosimetry can be accurately calculated for primary brain cancer patients using the pseudo-CT, thus allowing radiation treatment planning using MRI only. The IGRT treatments planned using qMRI will be compared to those planned conventionally.

The second part of the study (treatment monitoring) aims to evaluate the ability of qMRI techniques to provide clinical information such as distinguishing between progression and pseudo-progression, assessing treatment effectiveness or prognosis. The hypothesis is that qMRI can provide increased sensitivity to biological changes in tumors associated with disease progression over conventional (T1- or T2-weighted) MRI. The reasoning is that by providing quantitative, rather than weighted, images, direct numerical comparisons can be made between images acquired at different time points or at different centres. With traditional MRI, only limited, qualitative comparisons of tumor morphology or relative intensity within the same image can be made. Therefore, 3 or more follow-up MRI scans will also be acquired 3, 6 and 12 months after treatment and at recurrence, transformation, or pseudoprogression to monitor the effectiveness of the treatment.

These techniques will be tested on primary brain cancer patients undergoing IGRT, and the following data will be required:

1. the patient's IGRT treatment plan, as well as the planning CT and MRI datasets, and
2. additional scanning sessions approximately 45 minutes in duration to acquire MRIs of the patient with the new techniques at 3T. One of the sessions is prior to the beginning of the course of radiation therapy (first part of the study) and the remaining are after the completion of their radiation treatment (second part of the study).

Traditional treatment and follow-up care are unchanged.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Competent to sign informed consent.
* Diagnosed with primary tumor of the brain.
* Undergoing IGRT.
* Willing to participate in initial and follow up scan(s).
* Can lie supine in the MRI scanner for a period of about 45 minutes.
* Has signed informed consent.

Exclusion Criteria:

* Pregnancy.
* Contraindications to MRI (e.g., pacemakers, magnetic implants, metal in eye, claustrophobia).
* Has metallic implants in regions of interest (dental braces are okay).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Comparisons of radiation treatment plans by means of tumor control probabilities calculated from dose-volume histograms | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No